| HM-TRIA-102 Statistical | Analysis Plan | |
|---|---|---|
| | Statistical Ana | lysis Plan |
| | Protocol HM-T | |
| | tudy to Evaluate the Safety, and the safety, and the safety of Multiple Doses of HM | |
| | Phase | I |
| | | 1 |
| Prepared by: | | _ |
| Version: | Final | |

March 23, 2020

Date:

| HM-TRIA-102 Statistical Analysis Plan | |
|---|---|
| The Tree 102 Statistical Finallysis Flair | |
| Statistical Ar | nalysis Plan |
| Protocol HM | -TRIA-102 |
| A Phase 1 Study to Evaluate the Safety | y, Tolerability, Pharmacokinetics and |
| Pharmacodynamics of Multiple Doses of H | IM15211 in Obese Subjects with NAFLD |
| Phas | se I |
| Original Protocol: | 27 C 2010 |
| Version 1.0:<br>Version 2.0: | |
| Version 3:0:<br>Version 4.0: | 13-Feb-2019<br>09-Apr-2019 |
| Version 5.0: | - |
| This Statistical Analysis Plan has been reviewed a | and approved by: |
| · | |
| | Date: |



### **Table of Contents**

| 1. | Intr | oduction | 9 |
|---|---|---|---|
| 2. | Stu | dy Overview | 9 |
| | 2.1. | Study Design | 9 |
| | 2.2. | Randomization and Blinding | 11 |
| | 2.3. | Sample Size and Power | 11 |
| | 2.4. | Study Procedures and Visit Structure | 11 |
| 3. | Stu | dy Objectives | 11 |
| | 3.1. | Primary Objectives and Endpoints | 11 |
| | 3.1. | 1. Safety and Tolerability of HM15211 | 11 |
| | 3.1. | 2. Pharmacokinetics of HM15211 | 12 |
| | 3.1. | 3. Pharmacodynamics of HM15211 | 12 |
| | 3.2. | Exploratory Objectives and Endpoints | 12 |
| 4. | Ana | alysis Sets | 13 |
| | 4.1. | Safety Set | 13 |
| | 4.2. | Pharmacokinetic Analysis Set. | 13 |
| | 4.3. | Pharmacodynamic Analysis Set | 14 |
| 5. | Stu | dy Subjects | 14 |
| | 5.1. | Subject Disposition | 14 |
| | 5.2. | Demographic and Baseline Characteristics | 14 |
| | 5.3. | Medical History | 14 |
| | 5.4. | Subject Eligibility and Withdrawal Criteria | 14 |
| | 5.5. | Exposure | 14 |
| | 5.6. | Concomitant Medication | 15 |
| | 5.7. | Protocol Deviations | 15 |
| 6. | Sta | istical Methods of Analysis | 15 |
| | 6.1. | General Considerations | 15 |
| | 6.1. | 1. Statistical Notation and Presentation | 15 |
| | 6.1.<br>Obs | 2. Handling of Multiple Observations, Missing Observations or Out of Window servations | 16 |
| | 6.1. | 3. Handling of Missing or Partial Dates | 16 |
| | 6.1. | | |



| | 6.1.5. | Study Baseline | 18 |
|----|-----------|-------------------------------------------------------|----|
| 6. | 2. Pha | rmacokinetic Analyses | 18 |
| | 6.2.1. | PK Concentration | 18 |
| | 6.2.2. | PK Parameters | 18 |
| | 6.2.3. | Dose Proportionality | 19 |
| 6. | 3. Pha | rmacodynamic Analyses | 20 |
| | 6.3.1. | MRI-PDFF | 20 |
| 6. | 4. Exp | oloratory Analyses | 20 |
| | 6.4.1. | Incretins Secretion | 20 |
| | 6.4.2. | Body Weight, Body Mass Index, and Waist Circumference | 20 |
| | 6.4.3. | Serum Lipid Profile and Particles | 20 |
| | 6.4.4. | Amino Acids | 21 |
| | 6.4.5. | Inflammatory Marker | 21 |
| | 6.4.6. | Bone Metabolism | 21 |
| | 6.4.7. | Glucose Metabolism | 21 |
| | 6.4.8. | Ketone Bodies | 21 |
| | 6.4.9. | Liver Steatosis and Liver Stiffness | 21 |
| | 6.4.10. | Visceral Fat Volume | 22 |
| 6. | 5. Saf | ety Analyses | 22 |
| | 6.5.1. | Adverse Events | 22 |
| | 6.5.2. | Clinical Laboratory Assessments | 22 |
| | 6.5.3. | Immunogenicity | 22 |
| | 6.5.4. | Physical Examination | 23 |
| | 6.5.5. | Vital Signs | 23 |
| | 6.5.6. | 24-Hour Ambulatory Blood Pressure Monitoring | 23 |
| | 6.5.7. | 24-Hour Holter ECG | 23 |
| | 6.5.8. | 12-Lead Electrocardiograms | 23 |
| | 6.5.9. | Injection Site Reactions | 23 |
| 7. | Interim | Analysis | 24 |
| 8. | Statistic | al Software | 24 |
| 9. | Change | s to the Planned Analyses from Protocol | 24 |

| НМ-7 | RIA-102 Statistical Analysis Plan | |
|------|-----------------------------------|----|
| 10. | References | 24 |
| 11. | Appendix | 25 |



### **List of In-Text Tables and Figures**

| Table 1: Treatment Allocation and Dose Escalation (NAFLD) | 10 |
|-----------------------------------------------------------------|-----|
| Table 2: Schedule of Events, Cohorts 1-1 and 1-2 | 25 |
| Table 3: Schedule of Events, Cohorts 1-3 (not including Day 82) | 28 |
| Table 4: Schedule of Events, Cohorts 1-3 (including Day 82) | 31 |
| Table 5: Schedule of Events, Cohorts 1-4 | |
| Table 6: Schedule of Events, Cohorts 1-5 and up | 37 |
| Table 7: PK Sampling Schedule for cohorts 1-1 and 1-2 | |
| Table 8: PK Sampling Schedule starting from cohort 1-3 | |
| | 4.0 |
| Figure 1: Dose Escalation Schematic | 10 |



### **List of Abbreviations**

| List of Abbreviation | ons |
|---|---|
| Abbreviation | <b>Definition of Term</b> |
| obs | observed |
| _pred | predicted |
| ADAbs | Anti-drug antibodies |
| Adj_RSq | Adjusted r squared |
| AE | Adverse event |
| ANCOVA | Analysis of Covariance |
| anti-PEG | Anti-polyethylene glycol antibodies |
| ATC | Anatomic Therapeutic Chemistry |
| AUC | Area under the concentration-time curve |
| AUC0-168h SS | Area under the concentration-time curve for HM15211 during steady state |
| BLQ | Below the limit of quantitation |
| BMI | Body mass index |
| BP | Blood pressure |
| CAP | Controlled attenuation parameter |
| CI | Confidence interval |
| CL/F | Apparent clearance |
| Cmax | Maximum concentration |
| CSR | Clinical study report |
| Ctrough | Trough serum concentration |
| CTX-1 | Carboxy-terminal crosslinked telopeptide of type 1 collagen |
| CV | Cardiovascular |
| CV% | Coefficient of variation |
| ECG | Electrocardiogram |
| FFA | Free fatty acid |
| FGF21 | Fibroblast growth factor 21 |
| FPG | Fasting plasma glucose |
| GCG | Glucagon |
| GI | Gastrointestinal |
| GIP | Gastric inhibitory peptide |
| GLP-1 | Glucagon like peptide-1 |
| HA | Hyaluronic acid |
| HDL | High-density lipid |
| HDL-C | High-density lipid cholesterol content |
| HDL-P | High-density lipid particles |
| HR | Heart rate |
| IP | Investigational product |
| IWRS | Interactive Web Response System |
| kel | Apparent elimination constant |
| LDL | Low-density lipid |
| LDL-C | Low-density lipid cholesterol content |
| | * * |



| Abbreviation | Definition of Term |
|---|---|
| LDL-P | Low-density lipid particles |
| LLOQ | Lower limit of quantitation |
| LS | Least squares |
| LSM | Liver stiffness measurements |
| max | maximum |
| MedDRA | Medical dictionary for regulatory activities |
| min | minimum |
| MRI-PDFF | Magnetic resonance imaging-estimated proton density fat fraction |
| n | sample size |
| nAbs | Neutralizing antibodies |
| NAFLD | Non-alcoholic fatty liver disease |
| NCA | Non-compartmental analysis |
| NN | Normal to normal R-R intervals |
| OC | Osteocalcin |
| $P_1NP$ | Procollagen type 1 N-terminal propeptide |
| PD | Pharmacodynamics |
| PE | Physical examination |
| PK | Pharmacokinetics |
| PT | Preferred term |
| QTcF | Fridericia's corrected QT interval |
| $R_{dnm}$ | Ratio of the dose normalized geometric means |
| SAP | Statistical analysis plan |
| SC | Subcutaneous |
| SD | Standard deviation |
| SDANN | Standard deviation of the 5-minute average NN interval |
| SDNN index | Mean of standard deviations of all NN intervals for all 5 min |
| | segments of the entire recording. |
| SE | Standard error |
| SOC | System organ class |
| t1/2 | Half-life |
| TEAE | Treatment-emergent adverse event |
| Tmax | Time to maximum concentration |
| TSH | Thyroid stimulating hormone |
| VCTE | Vibration controlled transient elastography |
| VLDL | Very low-density lipid |
| VLDL-C | Very low-density lipid cholesterol content |
| VLDL-P | Very low-density lipid particles |
| Vz/F | Apparent volume of distribution at terminal |
| WHO DDE | World Health Organization drug dictionary enhanced |



### 1. Introduction

This document describes the statistical methods and data presentation in the analysis and summary of the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of HM15211 with Placebo as comparator in obese subjects with non-alcoholic fatty liver disease (NAFLD). This statistical analysis plan (SAP) was developed based on Hanmi Pharmaceutical Protocol HM-TRIA-102 (version 5.0 dated 02Jul2019).

This SAP will be finalized prior to data analyses and before database lock. Any major differences between the statistical methods provided in the clinical study protocol and this SAP will be explained herein. Any major changes and deviations from this SAP to the final data analysis must be substantiated by sound statistical rationale and fully documented in the final clinical study report (CSR).

### 2. Study Overview

### 2.1. Study Design

This is a randomized, placebo-controlled, multiple-ascending dose study to investigate the safety, tolerability, PK, and PD of subcutaneous (SC) administration of HM15211.

This study will be single-blind and conducted in up to 6 cohorts comprising a total of up to 72 obese subjects with NAFLD. Each cohort will enroll subjects to ensure that at least 12 subjects per cohort will complete the study. Subjects will be randomized to investigational product (IP) or placebo in a 3:1 ratio via an Interactive Web Response System (IWRS). Per cohort (n=12 subjects), 9 subjects will be randomized to HM15211 and 3 subjects to placebo. Cohorts may partially overlap after at least 9 subjects have completed 2-4 weeks of treatment (2 weeks of treatment is reached at Visit week 3) and a dose escalation decision has been made. Study drug will be administered weekly over a period of 12 weeks.

Based on the safety and available PK and PD data of each cohort, and following a safety review and dose escalation meeting between the investigator and the sponsor, dose escalation to the next cohort may proceed. Cohorts will start in sequential order but may overlap partially during execution. Replacement of dropouts and withdrawals may take place.

Each subject will undergo a screening visit, 2 in-house/ treatment periods and multiple outpatient visits. A final follow-up visit that will conclude subject study participation.

The duration of participation in this study including Screening, Treatment and Follow-up will be approximately 23 weeks for each subject including 12 weeks of treatment period.



**Table 1: Treatment Allocation and Dose Escalation (NAFLD)** 

| Cohorts | Number of Subjects | Treatment |
|------------|--------------------|--------------------|
| Cohort 1.1 | N=9 | HM15211 0.01 mg/kg |
| Cohort 1-1 | N=3 | Matching Placebo |
| Cohort 1-2 | N=9 | HM15211 0.02 mg/kg |
| Conort 1-2 | N=3 | Matching Placebo |
| | N=9 | HM15211 0.04 mg/kg |
| Cohort 1-3 | N=3 | Matching Placebo |
| Cohort 1-4 | N=9 | HM15211 0.06 mg/kg |
| Conort 1-4 | N=3 | Matching Placebo |
| Cohort 1-5 | N=9 | HM15211 0.08 mg/kg |
| Conort 1-5 | N=3 | Matching Placebo |
| Cohout 1.6 | N=9 | HM15211 0.12 mg/kg |
| Cohort 1-6 | N=3 | Matching Placebo |

Additional cohorts may be added if necessary, to provide sufficient data. Proposed doses for cohort 1-2 and 1-3 and 1-4 may be adjusted but will not exceed the doses stated in the table.

**Figure 1: Dose Escalation Schematic** 





### 2.2. Randomization and Blinding

Subjects who meet all inclusion and exclusion criteria or check-in criteria will be assigned a subject randomization number via an IWRS. The system will randomize in a 3:1 ratio to HM15211 or placebo. Randomization will continue until a total of up to 72 subjects have completed the study (or until 12 subjects per cohort have completed the study). If a subject fails to start dosing, or if a subject can't be randomized, the reason will be entered into the screening disposition page. The IWRS must be notified within 2 days that the subject was not randomized. In the event of an emergency, e.g. when it becomes necessary for the investigator to know which study drug the subject is taking, the subject code can be broken by the investigator, preferably after consultation with the medical monitor. Emergency code breaks can be performed using the IWRS, see section 8.7 in the protocol. As the study is single-blind, subjects and the clinical staff caring for the subjects are blinded to treatment. Staff involved in the data management, statistical analyses and staff from Pharmaceutical Services who are responsible for preparing the IP, will be unblinded. Unblinded staff will not be involved in the subjects' care.

After all subjects in one cohort have completed the Follow-up Visit, necessary steps to start with the data analysis may be taken. Data may be unblinded and data analysis for the completed cohort may start.

### 2.3. Sample Size and Power

Due to the exploratory nature of this study, a sample size of 12 subjects per cohort is empirically determined and consistent with typical sample sizes used for similar studies to assess PK and safety data.

### 2.4. Study Procedures and Visit Structure

In the appendix, Tables 2-6 describe the procedures and visit structure for this study for all Cohorts; Tables 7 and 8 describe the PK sampling schedules; the schedule of events and PK sampling schedules for each cohort can also be found in the clinical trial protocol.

### 3. Study Objectives

### 3.1. Primary Objectives and Endpoints

### 3.1.1. Safety and Tolerability of HM15211

To assess safety and tolerability of HM15211 after administration of multiple subcutaneous doses in obese subjects with NAFLD by:

- Incidence of adverse events (AEs) (cardiovascular [CV] events, rash/inflammatory dermatitis and other skin disorders, gastrointestinal [GI] events, and gall stone formation [cholelithiasis] will be managed following separate AE guidance document).
- Incidence of clinical lab abnormalities (including serum amylase, serum lipase, coagulation, thyroid stimulating hormone (TSH), serum calcitonin)



- Immunogenicity (Anti-drug antibodies [ADAbs], neutralizing antibodies [nAbs], antipolyethylene glycol antibodies [anti-PEG])
- Incidence and severity of clinical findings on physical examination
- Change from baseline in vital signs (blood pressure [BP], heart rate [HR], respiratory rate, and temperature]);
  - BP assessed by 24-hour ambulatory blood pressure monitoring (ABPM); HR assessed by 24-hour ambulatory electrocardiography monitoring (Holter ECG;
  - central reader)
- Change from baseline in 12-lead ECG parameters; the primary ECG endpoint will be QTcF
- Injection site reactions.

### 3.1.2. Pharmacokinetics of HM15211

To assess the pharmacokinetic (PK) profile of HM15211 after administration of multiple SC doses in obese subjects with NAFLD by, but not limited to:

- Maximum concentration (C<sub>max</sub>)
- Time to reach Cmax (t<sub>max</sub>)
- Trough serum concentration (C<sub>trough</sub>)
- Area under the concentration-time curve (AUC), eg, AUC<sub>0-t</sub> at steady state
- Terminal elimination rate constant (kel)
- Terminal half-life  $(t_{1/2})$
- Apparent clearance (CL/F)
- Apparent volume of distribution (Vz/F)

### 3.1.3. Pharmacodynamics of HM15211

To assess a reduction of liver fat after administration of multiple doses in obese subjects with NAFLD by:

• Absolute and % changes of fat on magnetic resonance imaging-estimated proton density fat fraction (MRI-PDFF)

### 3.2. Exploratory Objectives and Endpoints

To assess additional pharmacodynamic properties of HM15211 after multiple SC doses in comparison to placebo by:

- Incretins/ metabolic hormones
  - o Glucagon-like peptide-1 (GLP-1)
  - o Gastric inhibitory peptide (GIP)
  - o Glucagon
  - o Fibroblast growth factor 21 (FGF21)
  - o Leptin

| | | _ |
|----------------------|-------------------|---|
| HM-TRIA-102 Statisti | cal Analysis Plan | |

- Body weight and body mass index (BMI)
- Waist circumference
- Serum lipid profile and particles
  - o Total cholesterol
  - o Low-density lipoprotein (LDL): LDL-C, LDL-P (particles)
  - o High-density lipoprotein (HDL): HDL-C, HDL-P (particles)
  - o Very low-density lipoprotein (VLDL): VLDL-C, VLDL-P (particles)
  - o Triglycerides
  - o Free Fatty Acids (FFAs)
- Amino acid profile
- Inflammatory marker
  - o Adiponectin
- Bone metabolism parameters
  - o Fasting carboxy-terminal crosslinked telopeptide of type 1 collagen (CTX-1)
  - o Osteocalcin (OC)
  - o Procollagen type 1 N-terminal propeptide (P1NP)
- Glucose metabolism parameters:
  - o Fasting plasma glucose (FPG)
  - o Fasting insulin, fasting C-peptide
  - o HbA1c
- Ketone bodies
  - Beta-hydroxybutyrate
- Changes in liver steatosis and liver stiffness assessed by FibroScan® (VCTE), determined as absolute and percent change from baseline in controlled attenuation parameter (CAP) and liver stiffness measurements (LSM) (For Cohort 4 and 5)
- Changes in visceral fat volume, determined by absolute and relative percent change assessed by MRI imaging. (Will no longer be performed)

### 4. Analysis Sets

### 4.1. Safety Set

The Safety analysis set will include all subjects who received study medication (HM15211 or Placebo). The Safety analysis set will be used for demographic, baseline characteristics and safety summaries.

### 4.2. Pharmacokinetic Analysis Set

The PK analysis set will include all subjects who received HM15211 with evaluable PK data appropriate for the evaluation of interest (without important protocol deviations or violations that would have an impact on the absorption, distribution, metabolism, or excretion of HM15211). PK analysis set will be used for analysis of PK endpoints.



### 4.3. Pharmacodynamic Analysis Set

The PD analysis set will include all subjects who received HM15211 or placebo with evaluable PD data appropriate for the evaluation of interest (without important protocol deviations or violations that would have an impact on the PD of HM15211). PD analysis set will be used for analysis of PD endpoints.

### 5. Study Subjects

Study subject data will be summarized by treatment and treatment overall, with pooled placebo using the Safety Set.

### 5.1. Subject Disposition

Subject disposition will be summarized for the Safety Set. Summary tables will be presented.

### 5.2. Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized descriptively for all subjects in the Safety Set. Demographic and baseline characteristics include, but are not limited to: age, sex, ethnicity, race, body weight, height, body mass index, smoking status at Screening, alcohol use at Screening, VCTE, Liver Fat via MRI-PDFF, CAP and LSM by FibroScan®, HbA1c, c-peptide, insulin, fasting plasma glucose, total cholesterol, cholesterol and particles of HDL, LDL, and VLDL, triglycerides, Free Fatty Acids, creatinine, bilirubin, ALT, AST, GGT, and incretins/metabolic hormones.

### 5.3. Medical History

Medical history is any significant medical condition or disease that is present at study start (signing of informed consent). The medical history recorded through clinically significant laboratory, electrocardiogram (ECG), or physical examination (PE) abnormalities noted at Screening examination will be listed.

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA, version 23.0) and summarized by System Organ Class (SOC) and Preferred Term (PT) for the Safety Set. Medical history will be listed.

### 5.4. Subject Eligibility and Withdrawal Criteria

Subject eligibility and subjects who meet withdrawal criteria will be presented in listings.

### 5.5. Exposure

Total study dose administrated (mg/kg) and number of administration by visit and overall will be summarized by treatment and treatment overall, with pooled placebo. Study drug administration information will be listed.



### 5.6. Concomitant Medication

Concomitant medication is medication given in addition to the study medication (including overthe-counter medications, herbal medications, and vitamin supplements) administered between screening and follow-up. Medication will be categorized into the three following types:

- Prior concomitant medication is defined as any medications that start before the date of dosing of study medication and continue beyond that date.
- New concomitant medication is defined as any medications that start after the date of dosing of study medication, including those started in the follow-up period.
- Pre-treatment medication is defined as any non-study medication that stops before the date of dosing of study medication.

The WHO Drug Global version B3, March 2020) will be used to categorize the verbatim descriptions of medications into the Anatomic Therapeutic Chemistry (ATC) classification system. Each verbatim name will be classified by anatomical main group (ATC level 1), therapeutic subgroup (ATC level 2), pharmacological subgroup (ATC level 3), chemical subgroup (ATC level 4), and trade name.

The number and percentage of subjects receiving concomitant medications (including both prior and new concomitant medications) will be summarized by ATC classification (ATC level 2 and level 4) for the Safety Set. Pre-treatment medication administered during the study will only be listed.

### 5.7. Protocol Deviations

Protocol deviations may include the deviations from entry criteria, the study procedures, study medication intake/administration, or study restrictions, etc. Important protocol deviations will be identified prior to database lock and will be summarized for the Safety Set. Subjects with important protocol deviations that may impact the primary PK and PD endpoints will be excluded from the PK and PD Evaluable Sets. All deviations will be listed.

### 6. Statistical Methods of Analysis

### 6.1. General Considerations

PK, PD, and Safety analyses will be performed with the PK Evaluable Set, PD Evaluable Set, and Safety Set, respectively. All data collected during the study for Safety Set will be included in data listings.

### 6.1.1. Statistical Notation and Presentation

The continuous variables will be summarized by number of observations (n), mean, standard deviation (SD), median, minimum (min), and maximum (max). For categorical variables, the count and percentage of subjects in each category will be provided. For log-normal distributed data, geometric mean, standard error (SE) of the geometric mean, and coefficient of variation



(CV) will also be provided. The geometric mean is calculated as the exponential of the arithmetic mean calculated from data on a log scale. The CV is calculated as CV% = 100%\*  $sqrt(exp(\sigma^2) - 1)$ , where  $\sigma$  is the SD of the data on the natural log scale.

Minimum and maximum values will be rounded to the precision of the original value. Means, least squares (LS) means (if applicable), and medians will be rounded to 1 decimal place greater than the precision of the original value. SDs, SEs, and confidence intervals (CIs) will be rounded to 2 decimal places greater than the precision of the original value. Percentages for summarizing categorical data will be rounded to one decimal place. P-values, if needed, will be presented with 4 decimal places and values less than 0.0001 will be presented as <.0001.

All inferential statistical testing, if applicable, will be two-sided and conducted at the 0.05 significance level, unless specified otherwise. No multiplicity adjustment is planned for this study.

### 6.1.2. Handling of Multiple Observations, Missing Observations or Out of Window Observations

If there are multiple measurements within the same scheduled visit which are scheduled to be collected once at each visit and are recorded as triplicate 12-lead ECG's except the ECG at Screening, the average of the multiple measurements will be computed at each visit for all subjects and this averaged value will be used in all the analyses and summaries.

On scheduled visits with missing assessments, unscheduled assessments within the visit window, if available, may be used for analysis. Assessments collected during scheduled visits that are outside the visit window can be used for analysis. A footnote will be added to tables where unscheduled visits are used to impute missing scheduled visits.

For PK and PD data, if a blood sample was collected outside the protocol specified blood sampling time window, such data will still be included in data analysis, and the actual clock time will be used for PK and PD parameters calculations such as area under the curve (AUC).

All values, scheduled or unscheduled, will be presented in data listings.

### 6.1.3. Handling of Missing or Partial Dates

In cases of incomplete dates for adverse events (AEs) or non-study medications, the missing component(s) will be assumed as the most conservative value(s) possible. The imputation rule aims to capture AEs with missing start dates as treatment-emergent AEs (TEAEs) in a conservative manner with the following algorithms:

• If "day" is the only missing field, impute the "day" as the later one between the first day of the month and the dosing date if their "month" are the same.



- If "day" and "month" are the only missing fields, impute the "day" and "month" as the later one between January 1 of the year or the dosing date if the "year" is the same as the dose date.
- If "day", "month", and "year" are all missing, to be conservative, the event will be assumed to occur post-dose on the same day as the first dose administration day.

Concomitant medications with partial or missing start dates are assumed to have started prior to the dosing of the study medication. Non-study medications with missing or partial dates will be imputed similarly.

Date imputation will only be used for computational purposes; e.g., treatment-emergent status or identifying concomitant medications. Actual data values, as they appear in the clinical database, will be shown in the data listings.

### 6.1.4. Handling of Outliers and Unquantifiable Measurements

Prior to database lock, PK data will be reviewed by the principal investigator, pharmacokinetic scientists, consulting scientists, data management representatives, statisticians, and the sponsor to assess whether individual concentration values are inconsistent with other values from the same subject or if there are errors with the samples. The pharmacokineticist will provide input that will determine whether the sample result is plausible given the PK profile of the subject. Such values may be re-analyzed or may be removed from the analysis prior to calculation of PK parameters at the discretion of the pharmacokineticist. Determination of data points subject to re-analysis or removal from determination of PK parameters (i.e., implausible data) will be documented prior to database lock. Appropriate representatives will also review PK and PD parameter results and a determination of plausibility will be made. Individual subject results deemed implausible may be removed prior to summarization of PK and PD parameter results by treatment. Removal of individual subject PK/PD parameter results will be documented.

The following rules will be applied when blood samples are assayed as below the limit of quantitation (BLQ) or if individual concentration results are deemed implausible prior to database lock:

- For graphical presentations of the individual subject data: BLQ and values deemed implausible will not be displayed but will be flagged for reference and retained in the data as assayed.
- If any values are deemed implausible, final decisions and rationale will be documented in the pre-database lock meeting minutes.

For the calculation of summary statistics of concentrations or derivation of PK and PD parameters: values that are BLQ and values deemed implausible will be set to missing.



### 6.1.5. Study Baseline

Baseline will be defined as the last non-missing observation obtained prior to the administration of the study drug.

### 6.2. Pharmacokinetic Analyses

### 6.2.1. PK Concentration

Concentration of HM15211 will be summarized descriptively by treatment group. Line plots of HM15211 individual subject concentration overlaid with the mean concentration for each cohort will be plotted separately. In addition, a line plot of the HM15211 mean concentration by treatment group will be plotted.

### 6.2.2. PK Parameters

The following PK parameters will be derived using non-compartmental analysis and summarized by treatment group for the PK Analysis Set.

- Maximum concentration (C<sub>max</sub>) is defined as the maximum HM15211 concentration measured after SC dose. Will be calculated for Week 1 (1<sup>st</sup> dose) and Week 12 (12<sup>th</sup> dose):
  - o C<sub>max</sub> (Week 1)
  - o C<sub>max</sub> (Week 12)
- Time to reach  $C_{max}$  ( $T_{max}$ ) is defined as the time from initial injection to time of  $C_{max}$ . Will be calculated for Week 1 (1st dose) and Week 12 (12th dose):
  - o T<sub>max</sub> (Week 1)
  - o T<sub>max</sub> (Week 12)
- C<sub>trough</sub>, the trough serum concentration is defined as the minimum HM15211 concentration just prior to next dose administration. Will be calculated for Week 1 (pre 1<sup>st</sup> dose) and Week 12 (pre 12<sup>th</sup> dose):
  - o C<sub>trough</sub> pre-dose on Day 1 (Week 1)
  - o C<sub>trough</sub> pre-dose on Day 78 (Week 12)
- Area under the concentration-time curve for HM15211, AUC<sub>0-168h</sub> after 1<sup>st</sup> and 12<sup>th</sup> dosing (steady state), will be calculated by linear trapezoidal method.
  - o AUC<sub>0-168h</sub> (Week 1) and AUC<sub>0-inf</sub> (Week 1)
  - o AUC<sub>0-168h</sub> (Week 12)
- k<sub>el</sub>, first-order terminal elimination rate constant, calculated by linear regression of time vs. log concentration curve in the terminal phase. For k<sub>el</sub> to be acceptable, it shall be determined over a time interval equal to at least 1.5 x t½ k<sub>el</sub>, with at least three different time points in the terminal phase for the regression analysis, and the coefficient of



determination Adj\_RSq shall be  $\geq$ 0.8. If at least one of these three conditions is not fulfilled, the parameters depending on  $k_{el}$  (e.g., the terminal half-life t1/2  $k_{el}$ , CL and Vz) shall be flagged as not reliable if calculated and listed. They will generally be excluded from descriptive statistics and statistical testing procedures, unless otherwise judged by the pharmacokineticist in charge of PK analysis. Will be calculated for Week 1 (1st dose) and Week 12 (12th dose):

- o kel (Week 1)
- o kel (Week 12)
- Apparent terminal half-life t<sub>1/2</sub> will be determined from equation ln2/ k<sub>el</sub>. Will be calculated for Week 1 (1<sup>st</sup> dose) and Week 12 (12<sup>th</sup> dose).
  - $\circ$   $t_{1/2}$  (Week 1)
  - $\circ$   $t_{1/2}$  (Week 12)
- Apparent clearance divided by bioavailability (CL/F). Will be calculated for Week 1 (1<sup>st</sup> dose) and Week 12 (12<sup>th</sup> dose).
  - o CL/F (Week 1)
  - o CL/F (Week 12)
- Apparent volume of distribution at terminal phase divided by bioavailability (Vz/F). Will be calculated for Week 1 (1st dose) and Week 12 (12th dose).
  - o Vz/F (Week 1)
  - o Vz/F (Week 12)
- Accumulation ratio (AR). Will be calculated for Week 1 (1<sup>st</sup> dose) and Week 12 (12<sup>th</sup> dose).

Box plots of  $C_{max}$  and  $AUC_{0-168h\,SS}$  for each cohort may be generated.

### 6.2.3. Dose Proportionality

The power model will be used to analyze the dose proportionality in  $C_{max}$  and  $AUC_{0-168h SS}$  of HM15211. The estimate of the ratio of the dose normalized geometric means (mg/kg),  $R_{dnm}$ , and the corresponding 90% CI will be derived.

The power model is defined as follows:

$$log(PK_i) = \alpha + (\beta) * log(dose_i) + \mathcal{E}_i$$

Where

 $PK_i$  is the PK parameter ( $C_{max}$  or  $AUC_{0-168h}$ ) observation for the subject i.

 $\alpha$  is the population intercept.

 $\beta$  is the population slope.



 $\mathcal{E}_i$  is the random error;  $\mathcal{E}_i \sim N(0, \sigma_{\mathcal{E}}^2)$  and independent.

The assumption for the Power Model is that the underlying relationship between log(PK parameter) and log(dose) is linear. The dose proportionality corresponds to the ratio of dose-normalized geometric means ( $R_{dnm}$ ), which is defined as ratio of the predicted geometric mean of the highest dose relative to the predicted geometric mean of the lowest dose. The dose proportionality would be declared when the 90% CI for the  $R_{dnm}$  falls entirely within the limit of 0.8 to 1.25.

### 6.3. Pharmacodynamic Analyses

### **6.3.1.** MRI-PDFF

The observed values, change from baseline, and the percent change from baseline of liver fat on magnetic resonance imaging-estimated proton density fat fraction (MRI-PDFF) will be summarized descriptively by treatment group, visit, and time point.

A mixed model repeated measures analysis will be performed with the change from baseline in liver fat as the dependent variable, treatment group, analysis time point and the interaction between treatment group and analysis time point as factors, and the baseline of the dependent variable as a covariate. Repeated measures on each subject, at each visit week, will assume an unstructured covariance structure. If the model fails to converge, other covariance structures will be considered and selected based on model fit as determined by Akaike information criterion. The LS mean, SE of LS mean and 95% confidence interval will be presented by treatment group for each post baseline analysis time point. The LS mean difference from pooled placebo, SE of the LS mean difference from pooled placebo, and the 95% confidence interval will be presented by active treatment group for each post baseline analysis time point.

### 6.4. Exploratory Analyses

### 6.4.1. Incretins Secretion

Observed values and the change from baseline for parameters related to incretins secretion, such as GLP-1, GIP, GCG, FGF21, and leptin will be summarized descriptively by treatment group, visit, and time point. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.2. Body Weight, Body Mass Index, and Waist Circumference

The observed values, the change from baseline, and the percent change from baseline in body weight and waist circumference will be summarized by treatment group and visit. Observed values and change from baseline for BMI will be summarized similarly. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.3. Serum Lipid Profile and Particles

Observed values and the change from baseline for parameters related to lipid metabolism, such as total cholesterol, LDL-C, LDL-P, HDL-C, HDL-P, VLDL-C, VLDL-P, triglycerides, and



FFAs, will be summarized descriptively by treatment group and visit. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.4. Amino Acids

Observed values and the change from baseline for amino acids will be summarized descriptively by treatment group and visit. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.5. Inflammatory Marker

Observed values and the change from baseline for adiponectin will be summarized descriptively by treatment group and visit. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.6. Bone Metabolism

Observed values and the change from baseline for CTX-1, OC, and P<sub>1</sub>NP will be summarized descriptively by treatment group and visit. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.7. Glucose Metabolism

Observed values and the change from baseline for parameters related to glucose metabolism, such as FPG, fasting insulin, fasting C-peptide, and HbA1c will be summarized descriptively by treatment group, visit and time point. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.8. Ketone Bodies

Observed values and the change from baseline for beta-hydroxybutyrate will be summarized descriptively by treatment group and visit. MMRM analysis that will be specified similarly to the analysis of MRI-PDFF will be used.

### 6.4.9. Liver Steatosis and Liver Stiffness

Observed values and the absolute and percent change from baseline for CAP and LSM will be summarized descriptively by treatment group and visit. For Cohorts 4 and up, an analysis of covariance (ANCOVA) model with treatment as factor and baseline CAP (or LSM) value as a covariate will be performed to evaluate the change from baseline in CAP and LSM in each treatment group versus the pooled placebo group. The LS mean difference from pooled placebo, SE of the LS mean difference from pooled placebo, and the 95% confidence interval will be derived by treatment group for the single post-baseline visit. If data are not normally distributed based on the Shapiro-Wilks normality test, the Wilcoxon-Mann-Whitney test will be performed to analyze the change from baseline in CAP and LSM for each active treatment group versus the pooled placebo group. The Hodges-Lehmann estimator of the median and its 95% confidence interval will be provided.



### 6.4.10. Visceral Fat Volume

Visceral Fat Volume will no longer be collected or analyzed.

### 6.5. Safety Analyses

Safety data will be summarized by treatment, with pooled placebo. All safety data will be listed.

### 6.5.1. Adverse Events

Adverse events (AEs) will be coded using MedDRA, version 23.0. AEs will be summarized for the Safety Set.

AEs with onset on or after the date of informed consent but before the date of dosing of study medication will be considered pre-treatment AEs. Pre-treatment AE will be listed only.

AEs with onset date/time on or after receiving the dosing of study medication, or pre-existing AEs that increase severity on or after receiving the dosing of study medication will be considered as TEAE.

TEAEs will be summarized by SOC and PT, and by SOC, PT, and maximum severity by treatment group, with pooled placebo. TEAEs that are related to study medication per investigator's decision, TEAEs leading to study discontinuation, TEAEs that are serious (treatment-emergent SAEs) and adverse events of special interest (such as necrolytic migratory erythema, cholelithiasis and pancreatitis) will be summarized similarly.

AEs with missing severity will not be imputed. AEs with missing relationship will be imputed as related.

### 6.5.2. Clinical Laboratory Assessments

All hematology, clinical chemistry, and urinalysis results (including serum amylase, serum lipase, coagulation, thyroid stimulating hormone (TSH), serum calcitonin) will be summarized. Laboratory assessments that are outside of normal ranges and/or with potential clinical importance will be summarized and flagged in the listings. Shift tables of hematology, clinical chemistry, and urinalysis results will be generated to summarize the normal and abnormal (abnormal high and abnormal low) status changes from baseline.

### 6.5.3. Immunogenicity

Anti-drug antibodies (ADAbs, anti-HM15211 antibodies) will be summarized categorically, displaying the tier 1 (putative positive and negative) and tier 2 (positive and negative) tests by treatment group with positive tests further summarized by tier 3 absolute titer values and domain specificity. Tier 3 neutralizing antibody (nAbs) results will be summarized with ADAbs data in the same table.



In a separate table, anti-polyethylene glycol antibodies (anti-PEG) will be summarized categorically, displaying the screening result and specificity. The Anti-PEG specificity test will only be performed for samples where the titer increased more than 4 times compared to Day 1.

### 6.5.4. Physical Examination

The clinical findings on PE will have their incidence and severity listed.

### 6.5.5. Vital Signs

Observed vital sign values (blood pressure, heart rate, respiratory rate, and temperature) at each day and change from baseline at each post-baseline day will be summarized.

### 6.5.6. 24-Hour Ambulatory Blood Pressure Monitoring

Mean daytime (10:00 to 20:00) and nighttime (00:00-6:00) systolic and diastolic BP will be summarized for each day from Day -2 to Day 4 (Fagard 2008).

### 6.5.7. 24-Hour Holter ECG

Observed values from 24-Hour Holter ECG will be summarized by time point for each day from Day -1 to Day 4. Parameters calculated over the entire day such as mean HR, mean difference between day and night HR, mean NN intervals, pNN50, RMS SD, SDANN and SDNN index will be summarized by day.

Heart Rate Variability will be assessed by the following parameters:

- Percentage Greater than 50 msec (PRR\_GT50), aka pNN50, the percentage of successive differences in RR values greater than 50 milliseconds (can be increases or decreases) during the time period.
- RMS SD, the square root of the mean of the squares of successive differences between the RR values during the time period.
- Magid SD, also known as SDNN index, the average of five-minute period standard deviations of the RR intervals during the time period.
- Kleiger SD, also known as SDANN, standard deviation of all five-minute average RR intervals during the time period.

### 6.5.8. 12-Lead Electrocardiograms

Observed and change from baseline values of QTcF and other ECG parameters will be summarized. Status of 12-lead ECG parameters, normal, abnormal not clinically significant, and abnormal clinically significant, and their shifts from baseline will be summarized.

### 6.5.9. Injection Site Reactions

The number and percentage of subjects with any injection site reactions will be summarized by treatment group for the entire in-house period and by visit and time point within in-house period. The number and percentage of subjects with specific site reactions such as pain on palpation,



itching, erythema, edema, induration and other will be summarized by visit, time point, and Draize scale. In addition, diameter of affected areas will be summarized descriptively by visit and time point.

### 7. Interim Analysis

No interim analysis is planned.

### 8. Statistical Software

All statistical analyses will be performed using SAS® version 9.4. All PK and PD parameters will be derived with standard NCA methods using WinNonlin v5.2 or higher and/or SAS® version 9.4.

### 9. Changes to the Planned Analyses from Protocol

Visceral Fat Volume will no longer be collected or analyzed. Cohort 1-6 was not conducted.

### 10. References

Fagard RH, Celis H, Lutgarde T, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Daytime and nighttime blood pressure as predictors of death and cause-specific cardiovascular events in hypertension. *Hypertension*. 2008; **51**: 55-61.


HM-TRIA-102 Statistical Analysis Plan

### 11. Appendix

Table 2: Schedule of Events, Cohorts 1-1 and 1-2

| 7 8 9 10 11 43 50 57 64 71 77 78 X X X X X X X X X X X X X X |
|---|
| X X X X X X X X X X X X X X X X X X X |
| × |
| X X X |
| × |


HM-TRIA-102 Statistical Analysis Plan

| | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | , , | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| FU | Visit | 17 | 113 | <b>±2</b> | | | | | | X | X | X | | | | | | | | × | | | | | X | | | X | X | | | |
| ation | <b>Outpatient Visit</b> | 15 | 66 | <b>±</b> 2 | X | | | | | X | X | | | | | | | | | X | | | | | X | X | | X | X | | | |
| Elimination | Outps | 13 | 82 | | X | | | X | X | X | X | | | X | | X | X | X | X | X | | X | X | | X | X | | X | X | X | | |
| | | | 81 | | | | | | | | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| | iod 2 | 2 | 80 | | | | | | | | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| | In house Period 2 | 12 | 62 | | | | | | | | | | | | | | | | | X | | | | | | | | X | X | X | | |
| | In hou | | 28 | | X | | | | | X | X | | | | | | X | X | | × | | | | | X | X | | X | X | × | | |
| | | 1 | 77 | | | | | | | X | | | | | | | | | | × | | | | | | | | X | X | × | | |
| | | 11 | 71 | | | | | | | X | | | | | | | | | | X | | | | | | | | X | X | × | | |
| | | 10 | 64 | | | | | | | X | | | | | | | | | | × | | | | | | | | X | X | × | | |
| | | 6 | 57 | | × | | | X | | × | X | | | × | | × | × | × | × | × | | X | X | | X | | | X | X | × | | |
| po | sit | ∞ | 20 | | | | | | | × | | | | | | | | | | × | | | | | X | X | | X | X | × | | |
| Perio | ent Vi | 7 | 43 | | | | | | | X | | | | | | | | | | × | | | | | | | | X | X | × | | |
| Treatment Period | Outpatient Visit | 9 | 36 | | × | | | | | × | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| Trea | Õ | S | 50 | | X | | | X | X | X | X | | | | | | × | × | X | × | | | | | X | | | X | × | × | | |
| | | | | 4 | 22 | | | | | | | × | | | | | | | | | | × | | | | | X | X | | X | × | × |
| | | 3 | 15 | | X | | | X | | × | X | | | | | | × | × | | × | | | | | X | | | X | × | × | | |
| | | 7 | 10 | | | | | | | | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| | | | <b>∞</b> | | × | | | | | × | X | | | | | | × | × | | × | | | | | X | | | X | × | × | | |
| | | | 2-7 | | | | | | | | | | | | | | | | | × | | | | | | | | X | X | × | | |
| | od 1 | | 4 | | | | | | | | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| | se Peri | 1 | 2-3 | | | X | | | | | | | | | | | | | | × | | | | | X | | | X | X | × | | |
| | In House Period 1 | | 1 | | × | | | X | X | X | X | | | X | | | X | X | × | × | | X | X | | X | X | | X | X | X <sub>9</sub> | | |
| | | | -1 | | | | | | | | | | | | | | | | | | | | | nts | | | | X | × | | | |
| Admin | | | -2 | | | | | | | | | | | | | | | | | | | | | sessme | | | | X | X | | | |
| ; | <br>= | | -3 | | | | | | | | | | | | | | | | | | | | | city As | | | | | | | | |
| Come | Screen | | -44 to -3 | | X | | X | X | X | X | X | X | ssments | | | X | | | | | | | | nnogeni | | | ts | X | X | | | |
| | | Week | Day | Visit Window | Hematology,<br>Chemistry,<br>Coagulation, Urinalysis | CRP <sup>10</sup> | Lipid Panel | Amylase, Lipase | Calcitonin | Body Weight <sup>12</sup> | BMI Calculation | Waist Circumference | Pharmacodynamic Assessments | Lipid Profile and | Particles | MRI-PDFF <sup>5</sup> | Amino Acid Panel | Incretins <sup>6</sup> | Bone Metabolism | Glucose Metabolism | Parameters <sup>7</sup> | Inflammatory<br>Biomarkers <sup>11</sup> | Ketone Bodies | Pharmacokinetic and Immunogenicity Assessments | PK Sampling <sup>8</sup> | Immunogenicity | Other Safety Assessments | Adverse Event | Concomitant<br>Medication | Injection Site<br>Tolerability | | |

<sup>1</sup>Confirmation of eligibility

<sup>2</sup>Serum pregnancy test only at screening, urine pregnancy tests at all other time points
<sup>3</sup>Measurements of vital signs on PK sampling days will follow the PK sampling schedule and should be measured prior to every PK sample.

<sup>4</sup>ECG at screening not triplicate. ECG measurements are to be collected on Day-2 and 77 before subjects are connected to the ABPM and on Day 5 and 82 after subject have been disconnected from ambulatory device.

Subjects will undergo an MRI-PDFF assessment during week 8, as close as possible to Day 57, but prior to the Day 57 (week 9) Dosing and during week 12, as close as possible to Day 85, but prior to

the Day 85 PK sampling (week 13). <sup>6</sup>All incretins will be collected at the same time points together with the PK sample collection.


|--|


HM-TRIA-102 Statistical Analysis Plan

Table 3: Schedule of Events, Cohorts 1-3 (not including Day 82)

| | Č | Admin | nin | | | | | | | | | Treatment Period | nent Pe | eriod | | | | | | | | | Elimin | Elimination | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | screen | | | In H | ouse P | In House Period 1 | | | | | | Out | Outpatient Visit | t Visit | | | | | In h | ouse P | In house Period 2 | 2 | Out | Outpatient Visit | /isit |
| Week | | | | | | 1 | | | 2 | 3 | 4 | 5 | 9 | 7 | H | 9 10 | | 11 | | | 12 | | 13 | 15 | 17 |
| Day | -44 to -3 | -2 | -1 | 1 | 2-3 | 3 4 | 2-7 | 8 | 10 | 15 | 22 | 50 | 36 4 | 43 5 | 50 5 | 57 64 | 71 | 77 | 28 | 42 | 80 | 81 | 82 | 66 | 113 |
| Visit Window | | | | | | | | | | | | | | | | | | | | | | | | ±2 | 7∓ |
| Confinement | | X | × | X | X | X | X | X | | | | | | | | | 4 | × | × | × | × | × | | | |
| Dosing | | | | X | | | | X | | X | X | X | X . | X | X | X | X | | X | | | | | | |
| Randomization | | | X | | | | | | | | | | | | | | | | | | | | | | |
| Screening Procedures | | | | | | | | | | | | | | | | | | | | | | | | | |
| Informed Consent | × | | | | L | | | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | × | $\mathbf{X}_1$ | | | | | | | | | | | | | | | | | | | | | | | |
| Criteria | À | | | | | + | + | 1 | | | | | $\dagger$ | $\dagger$ | + | | + | $\downarrow$ | $\downarrow$ | - | $\downarrow$ | $\downarrow$ | | | |
| Demography | X | | | | | + | 1 | $\downarrow$ | | | | | $\dagger$ | + | + | | 4 | 4 | 1 | $\downarrow$ | 4 | 1 | | | |
| Medical History/Prior<br>Medication | × | | | | | | | | | | | | | | | | | | | | | | | | |
| Smoking and Alcohol | X | | | | | | | | | | | | | | | | | | | | | | | | |
| History | | | | | | | | | | | | | - | | | | | 4 | | | | _ | | | |
| Height | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Waist Circumference | X | | | | | | | | | | | | | | | | | | | | | | X | | X |
| Estimated Glomerular<br>Filtration Rate (eGFR) | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Thyroid Function Test (TSH) | X | | | X | | | | | | | | X | | | 7 | X | | | | | | | X | | X |
| HBA1C | × | | | | | | | | | | | | | | | | | | | | | | × | | |
| FPG | X | | | | | | | | | | | | | $\vdash$ | | | Ц | | | | | | | | |
| Serum Insulin | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Alpha-2 Macroglobulin | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Viral Serology | X | | | | | | | | | | | | | | | | | | | | | | | | |
| VCTE (FibroScan) | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Check-in Criteria to Inhouse Period | | X | | | | | | | | | | | | | | | | X | | | | | | | |
| Pregnancy Test <sup>2</sup> | X | × | | | | | | | X | X | × | × | × | X | X | X | X | X | | | | | X | X | X |
| Urine Drug Screen &<br>Alcohol Breath Test | X | X | | | | | | | × | X | × | | × | | X | | X | | | | | | × | X | X |
| Safety and Exploratory Assessments | Assessments | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical Examination (PE) | X | | | | | | | | | | | | | | | | | | | | | | | | X |
| Abbreviated PE | | X | | | | | | | | X | | X | | | ^ | X | | X | | | | | X | X | |
| Vital Signs <sup>3</sup> | X | X | X | X | X | | X | X | X | X | X | X | | X | X | XX | X | X | X | X | X | X | X | X | X |
| 12-lead ECG | $X^4$ | $X^4$ | | | | X | | | | × | | × | × | | ~ | <b>~</b> | _ | X | | | | × | | | |
| Holter Monitoring | | | × | × | × | | | | | | | | | | | | - | | × | × | × | × | | | |
| ABPM | | × | × | × | × | | - | | | | | | $\dashv$ | $\dashv$ | | | $\dashv$ | × | × | × | × | × | | | |


HM-TRIA-102 Statistical Analysis Plan

| | Č | Admin | nin | | | | | | | | | Treatment Period | ent Pe | riod | | | | | | | | | Elimination | ation | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | | | In E | In House Period 1 | eriod 1 | | | | | | Outp | Outpatient Visit | Visit | | | | | In ho | In house Period | eriod 2 | | Outp | Outpatient Visit | 'isit |
| Week | | | | | | 1 | | | 2 | 3 | 4 | Н | 2 9 | | 6 8 | 10 | | 11 | | Ţ | 12 | | 13 | 15 | 17 |
| Day | -44 to -3 | -2 | -1 | 1 | 2-3 | 4 | 2-7 | 8 | 10 | 15 | 22 | 29 3 | 36 4 | 43 5 | 50 57 | 64 | 71 | 77 | 28 | 62 | 80 | 81 | <b>S8</b> | 66 | 113 |
| Visit Window | | | | | | | | | | | | | | | | | | | | | | | | ∓2 | <b>±</b> 2 |
| Hematology, | X | | | X | | | | X | | X | | X | X | | X | | | | X | | | | X | X | |
| Chemistry, | | | | | | | | | | | | | | | | | | | | | | | | | |
| Coagulation, Urinalysis | | | | | | | | | | | | | 1 | + | | | | | | | | | | | |
| $CRP^{10}$ | | | | | X | | | | | | | | | | | | | | | | | | | | |
| Lipid Panel | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Amylase, Lipase | × | | | × | | | | | | × | | × | | | × | | | | | | | | × | | |
| Calcitonin | × | | | × | | | | | | | | X | | | | | | | | | | | × | | |
| Body Weight <sup>12</sup> | X | | × | $X^{12}$ | | | | X | | X | X | X | $\mathbf{x} = \mathbf{x}$ | | XX | X | X | X | X | | | | X | X | X |
| BMI Calculation | X | | | X | | | | X | | X | | × | | | X | | | | X | | | | X | X | X |
| Pharmacodynamic Assessments | ssments | | | | | | | | | | | | | | | | | | | | | | | | |
| Lipid Profile and | | | | X | | | | | | | | | | | X | | | | | | | | X | | |
| Particles | | | | | | | | | | | | | | | | | | | | | | | | | |
| MRI-PDFF <sup>5</sup> | X | | | | | | | | | | | | | | X | | | | | | | | X | | |
| Amino Acid Panel | | | | X | | | | X | | X | | X | | | X | | | | X | | | | X | | |
| Incretins <sup>6</sup> | | | | X | | | | X | | X | | X | | | X | | | | X | | | | X | | |
| Bone Metabolism | | | | X | | | | | | | | X | | | X | | | | | | | | X | | |
| Parameters | | | | | | | | | | | | | | - | | | | | | | | | | | |
| Glucose Metabolism | | | | × | X | X | X | X | X | X | X | X | $\mathbf{x} \mid \mathbf{x}$ | | $\mathbf{x} \mid \mathbf{x}$ | X | X | X | × | X | X | X | X | X | X |
| Parameters' | | | | | | | | | | | 1 | | 1 | + | | | | | | | | | | | |
| Inflammatory<br>Biomarkers <sup>11</sup> | | | | × | | | | | | | | | | | × | | | | | | | | × | | |
| Ketone Bodies | | | | × | | | | | | | | | | - | × | | | | | | | | × | | |
| Pharmacokinetic and Immunogenicity Assessments | nunogenicity | Assessr | nents | | | | | | | | | | | | | | | | | | | | | | |
| PK Sampling <sup>8</sup> | | | | X | X | X | | X | X | X | X | X | X | ` | X | | | | X | X | X | X | X | X | X |
| Immunogenicity | | | | X | | | | | | | X | | | 7 | X | | | | X | | | | X | X | |
| Other Safety Assessments | ıts | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X | X | X | X | X | $\mathbf{X} \mid \mathbf{X}$ | | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant | X | X | X | X | X | X | X | X | X | X | X | X | $\mathbf{x} = \mathbf{x}$ | | X | X | X | X | X | X | X | X | X | X | X |
| Medication | | | | | | | | | | | | | - | - | | | | | | | | | | | |
| Injection Site<br>Tolerability | | | | × | × | × | × | × | × | × | × | × | × | | × | × | × | × | × | × | × | × | × | | |
| Confirmation of eligibility | hility | | | | | | | | | | | | - | - | | | _ | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Confirmation of eligibility
<sup>2</sup>Serum pregnancy test and 10 other time points
<sup>3</sup>Measurements of vital signs on PK sampling days will follow the PK sampling schedule and should be measured prior to every PK sample.
<sup>4</sup>ECG at screening not triplicate. ECG measurements are to be collected on Day-2 and 77 before subjects are connected to the ABPM and on Day 4 and 81 after subject have been disconnected from ambulatory device.

Subjects will undergo an MRI-PDFF assessment during week 8, as close as possible to Day 57, but prior to the Day 57 (week 9) Dosing and during week 12, as close as possible to Day 85, but prior to the Day 85 PK sampling (week 13).

 $<sup>^6</sup>$ All incretins will be collected at the same time points together with the PK sample collection.  $^7$ Subjects need to be in fasting condition for collection.

| | lycic Dlan |
|-----|---------------------------------------|
| | TM TPIA 102 Statistical Analysis Dlan |
| - [ | É |

Page 30 Confidential

<sup>&</sup>lt;sup>8</sup>PK sampling will follow the PK sampling schedule. Cohort 3 will start to collect additional PK sample with start of Day 78.

<sup>9</sup>Injection site will be inspected pre-dose, at 4 and 12-hour post-dose on Day 1. Assessment of injection site on the other dosing days at least 30 minutes post-dose, and then daily during the in-house

periods and at outpatient visits on non-dosing days in the morning, approximately at the time of the dosing on dosing days. <sup>10</sup>CRP only, on Day 3. CRP is also measured at SCR/D1/D8/D15/D29/D36/D57/D78/D85/D99 in chemistry panel.

<sup>&</sup>lt;sup>11</sup>Inflammatory biomarkers will be collected at the same time points together with the PK sample collection.

<sup>&</sup>lt;sup>12</sup>To be measured prior to dosing.

<sup>13</sup>Weight to be collected in the moming, fasting and post void. On all dosing days, weight should be measured pre-dose.


HM-TRIA-102 Statistical Analysis Plan

Table 4: Schedule of Events, Cohorts 1-3 (including Day 82)

| _ | Τ. | | 3 | _, | | | 1 | | | 1 | 1 | 1 | | | 1 | 7 | | | | | 7 | | | | | | | Τ | <u> </u> | | <u> </u> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| FU | VISIT | + | 1113 | <b>±</b> 2 | | | | | | | - | - | | | | $\downarrow$ | _ | X | | | _ | × | | | | | 1 | | | × | × | | × | | X |
| ation | Outpatient visit | 15 | 99 | ∓7 | | | | | | | | | | | | | | | | | | | | | | | | | | × | × | | L | × | × |
| Elimination | Out | 13 | 68 | | | | | | | | | | | | | | | X | | | | × | × | | | | | | | X | × | | | × | X |
| | | 460 | <sub>2</sub> 78 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| • | 7 D | 5 | 81 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | × |
| - | e rerio | 12 | 80 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| - | in nouse Period 2 | É | 6/. | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| | II | Ç. | 8/ | | X | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | × |
| | Ī. | | 11 | | X | | | | | | ĺ | | | | | | | | | | | | | | | | | | × | X | × | | | × | X |
| ľ | - ; | = = | 1/1 | | | X | | | | | Ì | | | | | | | | | | 1 | | | | | | | | | X | × | 1 | | | × |
| | 9 | 01 | 64 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | X | | | | X |
| | • | 6 | 2/2 | | | X | | | | | | | | | | | | | | | | × | | | | | | | | X | × | | | X | × |
| Treatment Period | ııs | × ( | 20 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | | | | × |
| ment l | Outpatient visit | 7 5 | 43 | | | X | | | | | | | | | | | | | | | | | | | | | | | | × | × | | | | × |
| Treat | urpati | 9 } | 30 | | | X | | | | | | | | | | | | | | | | | | | | | | | | × | × | | L | | × |
| | ) | v 8 | 67 | | | × | | | | | | | | | | | | | | | | × | | | | | | | | × | × | | | × | × |
| | , | + | 77 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | | | L | × |
| | , | ر<br>ب | cI | | | × | | | | | | | | | | | | | | | | | | | | | | | | × | × | | | × | × |
| | _, | 7 | 10 | | | | | | | | | | | | | | | | | | _ | | | | | | | | | × | × | | | | × |
| | L | + | × | | X | X | | | | | | | | | | | | | | | 4 | | | | | | - | | | | | | | - | × |
| | | ı | ,-b | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| 7 | 100L | , | 4 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | × |
| - | In House Period 1 | 1 | 5-7 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| | III | , | I | | X | × | | | | | | | | | | | | | | | | × | | | | | | | | | | | | | × |
| nin | | + | -1 | | X | | × | | Г | | Ī | T | | | | | | | | | | | | | | | T | | | | | | | T | × |
| Admin | ľ | , | 7- | | X | | | | | $\mathbf{X}_1$ | | | | | | | | | | | | | | | | | | | × | X | × | nts | | × | × |
| Screen | | 77.77 | -44 to -<br>3 | | | | | | X | X | ; | X | < | | X | | X | X | X | | | × | X | X | X | × | × | × | | X | × | Assessme | X | | X |
| | | ¥ | Day | Visit Window | Confinement | Dosing | Randomization | Screening Procedures | Informed Consent | Inclusion/Exclusion | Criteria | Demography | Medical<br>History/Dries | Medication | Smoking and | Alcohol History | Height | Waist Circumference | Estimated | Glomerular Filtration | Kate (eGFR) | Thyroid Function<br>Test (TSH) | HBAIC | FPG | Serum Insulin | Alpha-2 | Viral Serology | VCTE (FibroScan) | Check-in Criteria to<br>In-house Period | Pregnancy Test <sup>2</sup> | Urine Drug Screen &<br>Alcohol Breath Test | Safety and Exploratory Assessments | Physical Examination | Abbreviated PE | Vital Signs <sup>3</sup> |
| | / * * | We | Day | Vis | Con | Dos | Ran | Scr | Info | Incl | 15 | Der | Mig<br>H | Mec | Smo | Alc | Hei | Wai | Esti | gg. | Kat | Thy<br>Test | HB, | FPC | Ser | Alp | Vir | VC | Che<br>In-b | Preg | Urii | Saf | Phy | (PE | (PE)<br>Abbr |

| Plan |
|------------|
| lysis |
| Anal |
| tatistical |
| .102 S |
| -TRIA- |
| HM |

| | Screen | Admin | min | | | | | | | | | Tr | eatmer | Treatment Period | po | | | | | | | | | Elimination | ation | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | In H | In House Period 1 | eriod 1 | | | | | | Outp | Outpatient Visit | Visit | | | | | I | n pons | In house Period 2 | od 2 | | Outpo | <b>Outpatient Visit</b> | isit |
| Week | | | | | | 1 | | | 2 | 3 | 4 | S | 2 9 | 2 8 | 6 | 10 | | 11 | | | 12 | | | 13 | 15 | 17 |
| Day | -44 to - | -2 | -1 | 1 | 2-3 | 4 | 5-7 | ∞ | 10 | 15 | 22 | 29 3 | 36 4 | 43 50 | 57 | 64 | 71 | 77 | 78 | 62 | 08 | 81 | *28 | 85 | 66 | 113 |
| Visit Window | | | | | | | | | | | | | | | | | | | | | | | | | ±2 | ±2 |
| 12-lead ECG | $X^4$ | $X^4$ | | | | × | | | | × | | X | × | | × | | | $X^4$ | | | | | X | | | |
| Holter Monitoring | | | × | X | × | × | | | | | | | | | | | | | X | X | X | X | X | | | |
| ABPM | | X | X | X | X | X | | | | | | | | | | | | X | X | X | X | X | X | | | |
| Hematology,<br>Chemistry | X | | | X | | | | X | | X | | × | X | | X | | | | X | | | | | X | X | |
| Coagulation,<br>Urinalysis | | | | | | | | | | | | | | | | | | | | | | | | | | |
| CRP <sup>10</sup> | | | | | × | | | | | | | | - | | | | | | | | | | | | | |
| Lipid Panel | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Amylase, Lipase | X | | | X | | | | | | × | | × | | | × | | | | | | | | | × | | |
| Calcitonin | X | | | X | | | | | | | | × | | | | | | | | | | | | X | | |
| Body Weight <sup>12</sup> | X | | X | $X^{12}$ | | | | X | | X | X | X | X | XX | X | X | X | X | X | | | | | X | X | X |
| BMI Calculation | X | | | X | | | | X | | X | | X | | | X | | | | X | | | | | X | X | X |
| Pharmacodynamic Assessments | sessments | | | | | | | | | | | | | | | | | | | | | | | | | |
| Lipid Profile and | | | | X | | | | | | | | | | | × | | | | | | | | | X | | |
| Particles | | | | | | | | | | | | | | | | | _ | | | | J | | | | | |
| MRI-PDFF <sup>5</sup> | X | | | | | | | | | | | | | - | × | | | | | | | | | X | | |
| Amino Acid Panel | | | | X | | | | X | | × | | × | + | | × | | _ | | X | | | | | X | | |
| Incretins <sup>6</sup> | | | | X | | | | X | | X | | X | | | × | | | | X | | | | | X | | |
| Bone Metabolism | | | | X | | | | | | | | × | | | X | | | | | | | | | X | | |
| I alameters | | | | ** | 1 | - | - | \$ | ì | þ | ; | + | + | + | + | + | þ | • | ì | 4 | • | 4 | | * | 4 | * |
| Glucose Metabolism<br>Parameters <sup>7</sup> | | | | × | < | <u> </u> | <b>&lt;</b> | × | × | × | <u> </u> | <u> </u> | ~<br>< | х<br> | <u> </u> | <u> </u> | < | × | × | < | × | × | | <b>×</b> | × | <b>×</b> |
| Inflammatory | | | | X | | | | | | | | | | | × | | | | | | | | | X | | |
| Biomarkers <sup>11</sup> | | | | Λ | | | | | | | | | | | > | | | | | | | | | > | | |
| Netolic Boules | | | ] | ₹ . | | | | | | | | | + | $\left \right $ | < | | | | | | | | | < | | |
| Pharmacokinetic and Immunogenicity Assessments | Immunoge | nicity | Asses | sments | | ; | _ | ; | ; | ; | ; | - | | - | ŀ | | | | ; | ; | ; | ; | ; | ; | ; | ; |
| PK Sampling° | | | | X | × | × | | X | X | × | × | X | X | X | × | | | | X | X | X | X | X | X | X | X |
| Immunogenicity | | | | X | | _ | _ | _ | | | × | | $\dashv$ | × | | | _ | | × | | | | | X | X | |
| Other Safety Assessments | ents | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X | X | X | X | | $\dashv$ | X | | X | × | X | X | X | X | X | X | X | X | X |
| Concomitant | X | X | X | X | X | × | × | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | × | X | X | X |
| Medication | | Ţ | Ī | 623 | , | - | - | • | • | Þ | > | | + | + | + | + | • | <b>&gt;</b> | • | • | • | • | • | * | | |
| Injection Site<br>Tolerability | | | | X' | × | X | × | X | X | × | × | X | X | xx | X | × | × | X | X | X | X | X | × | X | | |
| <sup>1</sup> Confirmation of eligibility | sligibility | | | | | | | | | | | | | | | | | | | | | | | | | |

\*Confirmation of eligiousty

2Serum pregnancy test only at screening, urine pregnancy tests at all other time points

3Measurements of vital signs on PK sampling days will follow the PK sampling schedule and should be measured prior to every PK sample.

ECG at screening not triplicate. ECG measurements are to be collected on Day-2 and 77 before subjects are connected to the ABPM and on Day 5 and 82 after subject have been disconnected from ambulatory device.

to the Day 57 (week 9) Dosing and during week 8, as close as possible to Day 57, but prior to the Day 57 (week 9) Dosing and during week 12, as close as possible to Day 85, but prior to the Day 85 PK sampling (week 13).

All incretins will be collected at the same time points together with the PK sample collection.

<sup>7</sup>Subjects need to be in fasting condition for collection.

PK sampling will follow the PK sampling schedule. Cohort 3 will start to collect additional PK sample with start of Day 78.

<sup>9</sup>Injection site will be inspected pre-dose, at 4 and 12-hour post-dose on Day 1. Assessment of injection site on the other dosing days at least 30 minutes post-dose, and then daily during the in-house periods and at outpatient visits on non-dosing days in the morning, approximately at the time of the dosing on dosing days.

<sup>0</sup>CRP only, on Day 3. CRP is also measured at SCR/DI/D8/DI5/D29/D36/D57/D78/D85/D99 in chemistry panel.

<sup>11</sup>Inflammatory biomarkers will be collected at the same time points together with the PK sample collection.

<sup>2</sup>To be measured prior to dosing.

<sup>13</sup>Weight to be collected in the moming, fasting and post void. On all dosing days, weight should be measured pre-dose.

\*Day 82 is optional for subjects already participating in cohort 1-3.


HM-TRIA-102 Statistical Analysis Plan

Table 5: Schedule of Events, Cohorts 1-4

| lan | |
|---------|---|
| Ы | |
| . 5 | |
| Analys | |
| < | |
| 12 | |
| Patisti | |
| V. | |
| 2 | 1 |
| Ξ | |
| ď | • |
| _ | |
| 2 | |
| 5 | |
| 2 | |
| Ħ | |

| | | Adı | Admin | | | | | | | | | Tre | atment | Treatment Period | - | | | | | | | | | Elimination | tion | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | | | In H | In House Period 1 | eriod 1 | | | | | | Outpa | Outpatient Visit | /isit | | | | | I | house | In house Period | 2 | | Outpatient | + | Visit |
| Week | | | | | | 1 | | | 2 | 8 | 4 | 9 9 | 7 | ∞ | 6 | 10 | = | | | | 12 | | | 13 | 15 | 17 |
| Day | -44 to - | -2 | -1 | 1 | 2-3 | 4 | 5-7 | ∞ | 10 | | 22 2 | - | 6 43 | 9 | 57 | 64 | 71 | 77 | 8/ | 62 | 08 | 81 | 82 | 85 | 66 | 113 |
| Visit Window | | | | | | | | | | | | | | | | | | | | | | | | | ±2 | ∓2 |
| 12-lead ECG | $X^4$ | $X^4$ | | | | X | | | | X | | X | | | X | | | $X^4$ | | | | | X | | | |
| Holter Monitoring | | | X | X | X | X | | | | | | | | | | | | | X | X | X | X | X | | | |
| ABPM | | X | X | X | X | X | | | | | | | | | | | | X | X | X | X | X | X | | | |
| Hematology, | × | | | X | | | | × | | X | | X | | | × | | | | × | | | | | X | × | |
| Chemistry, | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Coagulation, | | | | | _ | | | | | | | | | | | | | | | | | | | | | |
| CPD10 | | | | | > | $\downarrow$ | $\downarrow$ | | | | | | + | $\downarrow$ | | | | $\dagger$ | $\dagger$ | | $\dagger$ | | | | | |
| I inid Danel | > | | | | • | - | | | | | | | + | - | | | T | $\dagger$ | | + | + | l | Ī | | | |
| Amvlase, Linase | × | | | × | | | | | | × | | × | | | × | | | | | | | | | × | | |
| Calcitonin | × | | | × | | | | | | 1 | | : × | $\vdash$ | | 1 | | T | T | | t | t | l | | × | | |
| Body Weight <sup>12</sup> | × | | × | $X^{12}$ | | L | | × | | × | × | X | × | × | × | × | × | × | × | | - | | | × | × | × |
| BMI Calculation | × | | | × | | | | × | | × | | | | | × | | | | × | | | | | × | × | × |
| Pharmacodynamic Assessments | sessments | | | | | | | | | | | | | | | | | | | | | | | | | |
| Lipid Profile and | | | L | × | | | | | | | | | L | L | × | | | | r | r | | H | | × | | |
| Particles | | | | | | | | | | | | | | | | | | | | | | | | | | |
| MRI-PDFF <sup>5</sup> | X | | | | | | | | | | | | | | X | | | | | | | | | X | | |
| Amino Acid Panel | | | | X | | | | X | | X | . 1 | X | | | × | | | | × | | | | | X | | |
| Incretins <sup>6</sup> | | | | X | | | | X | | X | . 1 | X | | | X | | | | X | | | | | X | | |
| Bone Metabolism | | | | X | | | | | | | 1 | X | | | × | | | | | | | | | X | | |
| Parameters | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Glucose Metabolism | | | | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | | × | × | × |
| Parameters' | | | | ļ | | | | | | | | | - | | ; | | | | 1 | | | | | ķ | | |
| Inflammatory<br>Biomarkers <sup>11</sup> | | | | × | | | | | | | | | | | × | | | | | | | | | × | | |
| Ketone Bodies | | | | X | | | | | | | | | | | × | | | | | | | | | X | | |
| Pharmacokinetic and Immunogenicity Assessments | Immunogo | enicity | Asses | sments | | | | | | | | | | | | | | | | | | | | | | |
| PK Sampling <sup>8</sup> | | | | X | X | X | | X | X | X | X | X | | X | X | | | | X | X | X | X | X | X | X | X |
| Immunogenicity | | | | X | | | | | | | X | | | X | | | | | X | | | | | X | X | |
| Other Safety Assessments | ents | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X | X | X | X | $\mathbf{x} \mid \mathbf{x}$ | X 3 | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant | X | X | × | X | X | × | X | X | × | × | × | X X | X . | × | × | X | × | × | × | X | × | × | X | X | X | X |
| Injection Site | | $oxed{\bot}$ | | X <sub>9</sub> | × | × | × | × | × | × | × | X | × | × | × | × | × | × | × | × | × | × | × | X | T | |
| Tolerability | | | | | : | ! | 1 | : | | : | | | | | ; | : | : | : | : | : | : | : | : | | | |
| <sup>1</sup> Confirmation of eligibility | sligibility | | | | | | | | | | | | | | | | | | | | | | | | | |

'Confirmation of eligibility

<sup>2</sup>Serum pregnancy test only at screening, urine pregnancy tests at all other time points

<sup>3</sup>Measurements of vital signs on PK sampling days will follow the PK sampling schedule and should be measured prior to every PK sample.


ECG at screening not triplicate. ECG measurements are to be collected on Day-2 and 77 before subjects are connected to the ABPM and on Day 5 and 82 after subject have been disconnected from

Subjects will undergo an MRL-PDFF assessment during week 8, as close as possible to Day 57, but prior to the Day 57 (week 9) Dosing and during week 12, as close as possible to Day 85, but prior to the Day 85 PK sampling (week 13).

<sup>6</sup>All incretins will be collected at the same time points together with the PK sample collection.

7Subjects need to be in fasting condition for collection.

<sup>8</sup>PK sampling will follow the PK sampling schedule.

Phjection site will be inspected pre-dose, at 4 and 12-hour post-dose on Day I. Assessment of injection site on the other dosing days at least 30 minutes post-dose, and then daily during the in-house

periods and at outpatient visits on non-dosing days in the morning, approximately at the time of the dosing on dosing days. <sup>10</sup>CRP only, on Day 3. CRP is also measured at SCR/D1/D8/D15/D29/D36/D57/D78/D85/D99 in chemistry panel.

<sup>13</sup>Weight to be collected in the moming, fasting and post void. On all dosing days, weight should be measured pre-dose. <sup>1</sup>Inflammatory biomarkers will be collected at the same time points together with the PK sample collection. <sup>12</sup>To be measured prior to dosing.


HM-TRIA-102 Statistical Analysis Plan

Table 6: Schedule of Events, Cohorts 1-5 and up

| | | | | | | | ı | | | I | | 1 | l | | Т | | 1 | | | | _ | | ı | <u> </u> | | | Т | Т | l | | г | _ | T | | П | $\neg$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| FU | Visit | 17 | 113 | ±2 | | | | | | | | | | | | | | X | | | | × | | | | | | | | X | × | | ļ | × | | X |
| ation | Outpatient Visit | 15 | 66 | <b>7</b> | | | | | | | | | | | | | | | | | | | | | | | | | | X | X | | | | X | X |
| Elimination | Outpa | 13 | 85 | | | | | | | | | | | | | | | X | | | | × | X | | | | | X | | X | X | | | | X | X |
| | | | 82 | | X | | | | | | | | | | Ī | | | | | | | | | | | | | | | | | | ŀ | | | X |
| | 2 | | 81 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | - | ŀ | | | X |
| | Period | 12 | 08 | | X | - | | | - | | | | | | | | | | | | | | | | | | | | | | | 1 | ŀ | | | X |
| | In house Period 2 | | 62 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | - | ŀ | | | X |
| | In | | - 28 | | X | X | | | - | | | | | | | | | | | | | | | | | | | | | | | 1 | ŀ | | | X |
| | | | 77 | | X | | | | - | | | | | | | | | | | | | | | | | | | | × | X | × | 1 | ŀ | | X | X |
| | | 11 | 71 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | - | ŀ | | | X |
| | | 10 | 64 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | | ŀ | | | X |
| | | 6 | 57 | | | X | | | | | | | | | | | | | | | | × | | | | | | | | X | × | 1 | ľ | | X | X |
| eriod | it | × | 20 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | 1 | ľ | | | X |
| Treatment Period | Outpatient Visit | 7 | 43 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | X | | | | | X |
| Freatr | ıtpatie | 9 | 36 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | | L | | | X |
| | 0 | w | 29 | | | × | | | | | | | | | | | | | | | | × | | | | | | | | X | × | | L | | × | X |
| | | 4 | 22 | | | X | | | | | | | | | | | | | | | | | | | | | | | | X | × | | L | | | X |
| | | 3 | 15 | | | × | | | | | | | | | | | | | | | | | | | | | | | | × | × | | | | × | X |
| | | 7 | 10 | | | | | | | | | | | | | | | | | | | | | | | | | | | X | × | | | | | X |
| | | | ∞ | | X | X | | | | | | | | | | | | | | | | | | | | | | | | | | | L | | | X |
| | | | 2-7 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | × |
| | iod 1 | | 4 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| | In House Period 1 | 1 | 2-3 | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X |
| | In Ho | | 1 | | X | X | | | | | | | | | | | | | | | | × | | | | | | | | | | | ľ | | | X |
| nin | | | 7 | | X | | × | | | | | | | | Ī | | | | | | | | | | | | T | | | | | 1 | ľ | | | X |
| Admin | | | -2 | | X | | | | | $\mathbf{X}_1$ | | | | | | | | | | | | | | | | | | | × | X | × | nts | - | | X | X |
| | naarac | | -44 to - | | | | | | × | X | | X | X | | • | × | X | X | X | | | × | X | X | X | X | × | × | | X | X | Assessme | The second | × | | X |
| | | | | | | | | edures | int | sion | | | | | 1 | | | rence | | ration | | u. | | | | | | an) | ia to | ì | en & | lest | TOT WELL | nation | | |
| | | Week | Day | Visit Window | Confinement | Dosing | Randomization | Screening Procedures | Informed Consent | Inclusion/Exclusion | Criteria | Demography | Medical | History/Prior<br>Medication | 1 | Smoking and<br>Alcohol History | Height | Waist Circumference | Estimated | Glomerular Filtration | Rate (eGFR) | Thyroid Function<br>Test (TSH) | HBAIC | FPG | Serum Insulin | Alpha-2 | Viral Serology | VCTE (FibroScan) | Check-in Criteria to<br>In-house Period | Pregnancy Test <sup>2</sup> | Urine Drug Screen & | Safety and Exploratory Assessments | Dancy and Lap | Physical Examination (PE) | Abbreviated PE | Vital Signs <sup>3</sup> |

HM-TRIA-102 Statistical Analysis Plan

| | ū | Admin | nin | | | | | | | | | Trea | ıtment | Treatment Period | | | | | | | | | E | Elimination | ion | FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | | | In Ho | In House Period | riod 1 | | | | | | Outpa | Outpatient Visit | isit | | | | | In ] | louse l | In house Period 2 | 2 | | Outpatient Visit | ent Vi | sit |
| Week | | | | | | 1 | | | 2 | 3 | 4 | 9 9 | 7 | 8 | 6 | 10 | 11 | | | | 12 | | | 13 | 15 | 17 |
| Day | -44 to - | -2 | -1 | 1 | 2-3 | 4 | 5-7 | ∞ | 10 | 15 2 | 22 2 | 29 36 | 5 43 | 20 | 57 | 49 | 71 | | - 82 | 8 62 | 80 81 | - | 83 | 85 | 66 | 113 |
| Visit Window | | | | | | | | | | | | | | | | | | | | | | | | | ∓2 | ±2 |
| 12-lead ECG | $X^4$ | $X^4$ | | | | X | | | | X | ` | X | | | X | | | $X^4$ | | | | ` | X | | | |
| Holter Monitoring | | | X | X | X | X | | | | | | | | | | | | | X | X | X X | | X | | | |
| ABPM | | X | X | X | X | X | | | | | | | | | | | | X | X | X | X X | | X | | | |
| Hematology,<br>Chemistry, | X | | | X | | | | X | | × | | x x | | | X | | | | × | | | | | × | X | |
| Coagulation, | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urinalysis | | | | | ì | | | | | | | | | $\prod$ | | 1 | | | | + | | | | | | |
| $\mathbb{C}\mathbf{RP}^{10}$ | | | | | X | | | | | | | | | | | | | | | | | | | | | |
| Lipid Panel | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Amylase, Lipase | X | | | X | | | | | | X | 7 | X | | | X | | | | | | | | | X | | |
| Calcitonin | X | | | X | | | | | | | ^ | X | | | | | | | | | | | | X | | |
| Body Weight <sup>12</sup> | X | | X | $X^{12}$ | | | | X | | X | X | $\mathbf{X} \mid \mathbf{X}$ | X | X | X | X | X | × | X | | | | | X | X | × |
| BMI Calculation | X | | | X | | | | X | | X | ^ | X | | | X | | | | X | | | | | X | X | × |
| Pharmacodynamic Assessments | sessments | | | | | | | | | | | | | | | | | | | | | | | | | |
| Lipid Profile and | | | | X | | | | | | | | | | | X | | | | | | | | | X | | |
| Particles | ì | | | | | | | | Ī | | | | - | $\prod$ | þ | T | | | | 1 | + | 1 | | | | |
| MKI/MKI-PDFF | X | | | | | | | | | | | | + | Ţ | X | 1 | 1 | | | $\dagger$ | 1 | | | X | | |
| Amino Acid Panel | | | | X | | | | × | | × | ~ | X | _ | | × | | | | × | $\dashv$ | 1 | | | X | | |
| Incretins <sup>6</sup> | | | | X | | | | X | | × | 7 | X | | | X | | | | X | | | | | X | | |
| Bone Metabolism | | | | × | | | | | | | | <b>×</b> | | | × | | | | | | | | | × | | |
| Parameters | | | | | | | | | | | | | $\dashv$ | | | | | | | | | | | | | |
| Glucose Metabolism | | | | × | X | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | | × | × | × |
| Parameters' | | | | > | | | | | | | | | + | | > | | | | | + | | | | > | | |
| Biomarkers <sup>11</sup> | | | | < | | | | | | | | | | | < | | | | | | | | | < | | |
| Ketone Bodies | | | | X | | | | | | | | | | | X | | | | | | | | | X | | |
| Pharmacokinetic and Immunogenicity Assessments | Immunoge | nicity | Asses | sments | | | | | | | | | | | | | | | | | | | | | | |
| PK Sampling <sup>8</sup> | | | | X | X | X | | X | X | X | X | X | | X | X | | | | X | X | X | | X | X | X | X |
| Immunogenicity | | | | X | | | | | | | X | | | X | | | | | X | | | | | X | X | |
| Other Safety Assessments | ents | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X | X | X | X | XX | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant | X | X | X | X | X | X | X | X | X | X | X | $\mathbf{X} \mid \mathbf{X}$ | X | X | X | X | X | X | X | X | X | X | × | X | X | × |
| Medication | | | | 0 | ì | ÷ | , | ; | ; | | + | | + | ; | ţ | ; | ; | + | +; | + | + | + | | ļ | † | T |
| Injection Site<br>Tolerability | | | | × | × | × | × | × | × | × | <u>~ </u> | <u>×</u> | × | × | × | × | × | × | × | × | <u>~</u><br>× | <u> </u> | <u> </u> | × | | |
| <sup>1</sup> Confirmation of eligibility | eligibility | | | | | | | | | | | | | | | | - | | | | | | | | | |

'Confirmation of eligibility
<sup>2</sup>Serum pregnancy test only at screening, urine pregnancy tests at all other time points
<sup>3</sup>Measurements of vital signs on PK sampling days will follow the PK sampling schedule and should be measured prior to every PK sample.


ECG at screening not triplicate. ECG measurements are to be collected on Day-2 and 77 before subjects are connected to the ABPM and on Day 5 and 82 after subject have been disconnected from ambulatory device.

undergo an MRI/MRI-PDFF assessment during week 8, as close as possible to Day 57, but prior to the Day 57 (week 9) Dosing and during week 12, as close as possible to Day 85, but prior to the Day 85 PK sampling (week 13).

All incretins will be collected at the same time points together with the PK sample collection.

'Subjects need to be in fasting condition for collection.

<sup>8</sup>PK sampling will follow the PK sampling schedule.

Phjection site will be inspected pre-dose, at 4 and 12-hour post-dose on Day I. Assessment of injection site on the other dosing days at least 30 minutes post-dose, and then daily during the in-house

periods and at outpatient visits on non-dosing days in the morning, approximately at the time of the dosing on dosing days. <sup>10</sup>CRP only, on Day 3. CRP is also measured at SCR/D1/D8/D15/D29/D36/D57/D78/D85/D99 in chemistry panel.

<sup>13</sup>Weight to be collected in the moming, fasting and post void. On all dosing days, weight should be measured pre-dose. <sup>1</sup>Inflammatory biomarkers will be collected at the same time points together with the PK sample collection. <sup>12</sup>To be measured prior to dosing.


Table 7: PK Sampling Schedule for cohorts 1-1 and 1-2

| | PK samplii | PK sampling schedule | |
|---|---|---|---|
| | | T. S. C. | Pre-dose 1st dosing |
| | | Day I | 8 h after 1st dosing |
| | Week 1 | Day 2 | 24 h after 1st dosing |
| | | Day 3 | 48 h after 1st dosing |
| | | Day 4 | 72 h after 1st dosing |
| | | Day 8 | Pre-dose 2 <sup>nd</sup> dosing |
| | Week 2 | Day 10 | 48 h after 2 <sup>nd</sup> dosing |
| | Week 3 | Day 15 | Pre-dose 3rd dosing |
| Treatment Period | Week 4 | Day 22 | Pre-dose 4th dosing |
| | Week 5 | Day 29 | Pre-dose 5 <sup>th</sup> dosing |
| | Week 6 | Day 36 | Pre-dose 6 <sup>th</sup> dosing |
| | Week 8 | Day 50 | Pre-dose 8 <sup>th</sup> dosing |
| | Week 9 | Day 57 | Pre-dose 9 <sup>th</sup> dosing |
| | | Des 78 | Pre-dose 12 <sup>th</sup> dosing |
| | Wooly 13 | Day /o | 8 h after 12 <sup>th</sup> dosing |
| | Week 12 | Day 80 | 48 h after 12 <sup>th</sup> dosing |
| | | Day 81 | 72 h after 12 <sup>th</sup> dosing |
| Flimination Donica (+2) | Week 13 | Day 85 | 168 h after 12 <sup>th</sup> dosing |
| | Week 15 | Day 99 | 504 h after 12 <sup>th</sup> dosing |
| $\mathrm{F/U}~(\pm 2)$ | Week 17 | Day 113 | 840 h after 12 <sup>th</sup> dosing |


Table 8: PK Sampling Schedule starting from cohort 1-3

| | PK sampli | PK sampling schedule | |
|---|---|---|---|
| | | | Pre-dose 1st dosing |
| | | Day 1 | 8 h after 1st dosing |
| | West | Day 2 | 24 h after 1st dosing |
| | week 1 | Day 3 | 48 h after 1st dosing |
| | | Day 4 | 72 h after 1st dosing |
| | | Day 5* | 96 h after 1st dosing |
| | C TO SIM | Day 8 | Pre-dose 2 <sup>nd</sup> dosing |
| | week 2 | Day 10 | 48 h after 2 <sup>nd</sup> dosing |
| | Week 3 | Day 15 | Pre-dose 3rd dosing |
| Treatment Period | Week 4 | Day 22 | Pre-dose 4 <sup>th</sup> dosing |
| | Week 5 | Day 29 | Pre-dose 5 <sup>th</sup> dosing |
| | Week 6 | Day 36 | Pre-dose 6 <sup>th</sup> dosing |
| | Week 8 | Day 50 | Pre-dose 8 <sup>th</sup> dosing |
| | Week 9 | Day 57 | Pre-dose 9th dosing |
| | | Doy 78 | Pre-dose 12th dosing |
| | | Day /8 | 8 h after 12 <sup>th</sup> dosing |
| | Week 12 | Day 80 | 48 h after 12 <sup>th</sup> dosing |
| | | Day 81 | 72 h after 12 <sup>th</sup> dosing |
| | | Day 82** | 96 h after 12 <sup>th</sup> dosing |
| Flimingtion Donied | Week 13 | Day 85 | 168 h after 12 <sup>th</sup> dosing |
| Emiliation reflot (±2) | Week 15 | Day 99 | 504 h after 12 <sup>th</sup> dosing |
| $\mathrm{F/U}~(\pm 2)$ | Week 17 | Day 113 | 840 h after 12 <sup>th</sup> dosing |
| | | • | 1 |

<sup>\*</sup>Sampling on Day 5 will start with Cohort 1-4 and will not be taken for cohort 1-3.


<sup>\*\*</sup>Sampling on Day 82 will be optional for cohort 1-3 but will be taken in cohort 1-4.